CLINICAL TRIAL: NCT01641848
Title: Limited Enrollment of the INBONE™ Total Ankle Prosthesis With Long Talar Stem
Brief Title: INBONE™ Total Ankle Prosthesis With Long Talar Stem
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of patient enrollment
Sponsor: Stryker Trauma and Extremities (Industry)
Collaborators: Orthopedic Foot and Ankle Center, Ohio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-SJA-002
Record Dates: First submitted 2011-06-03; First posted 2012-07-17 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2013-08

CONDITIONS: Arthritis; Infection of Total Ankle Joint Prosthesis
Keywords: Total Ankle Arthroplasty
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arthritic and injured ankles (Experimental): InBone TAA
  Interventions: Device: INBONE™ Total Ankle Prosthesis with Long Talar Stem

INTERVENTIONS:
Device: INBONE™ Total Ankle Prosthesis with Long Talar Stem — INBONE™ Total Ankle Prosthesis with Long Talar Stem when used with a Calcaneal Stem

SUMMARY:
The primary objective of this study is to collect preoperative, operative and postoperative clinical assessments of patients that qualify for surgical implantation of the INBONE™ Total Ankle Prosthesis.

DETAILED DESCRIPTION:
The FDA approved the "limited enrollment" registry to provide us with additional clinical data from which to design a pivotal IDE study. FDA has stated that their decision for this was based upon "adequate safety information" which was submitted to them as part of the original IDE submission. Therefore, the purpose of this "limited enrollment" registry study is to gather initial data on the device's performance, when used with a Calcaneal Stem.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has sufficient soft tissue and muscle strength to support stable, anatomic positioning and motion of arthroplasty components as determined by the investigator
2. Subject must have sufficient skin for wound coverage.
3. Subject demonstrates subtalar joint insufficiency as defined by any of the following:

(1)range of motion <50 percent of the contralateral, non-diseased side (2)pain during physical examination of the subtalar joint (3)fusion

AND

Subject demonstrates tibio-talar joint insufficiency as defined by any of the following:

1. end stage arthritis as determined by the investigator on plain radiographs
2. pain during physical examination of the tibio-talar joint
3. fusion
4. non-union
5. failed Total Ankle Replacement 4.Subject has Body Mass Index (BMI) < 40 5.Subject has sufficient calcaneal bone stock as determined by the investigator 6.Subject is able to or capable of providing consent to participate in the clinical investigation and has medical insurance to cover costs associated with their medical care or is willing to assume personal responsibility for costs 7.Subject agrees to comply with this protocol, including participating in required follow-up visits at the investigations site and completing study questionnaires

Exclusion Criteria:

1. Subject is skeletally immature and under 21 years of age
2. Subject has experienced local or systemic infection within the past twelve months
3. Subject has symptomatic ankle disease or has been treated operatively on the contralateral side
4. Subject has vascular and kidney insufficiencies
5. Subject is suspected to have neuropathy of the foot or ankle
6. Subject has impaired vascular circulation in the affected limb
7. Subject has skin condition that may impair wound healing
8. Subject has known allergy to cobalt, chromium, molybdenum, titanium, aluminum, vanadium, or nickel
9. Subjects on long term medications which may compromise bone stock (e.g. long term steroids, NSAIDS, etc., physicians discretion
10. Subject is unwilling or unable to comply with a rehabilitation program
11. Subject is known to be pregnant, a prisoner, mentally incompetent, and/or alcohol or drug abuser
12. Subject is currently participating in any investigational study not related to this study's preoperative and postoperative care.
13. Subject has rheumatoid arthritis (RA)
14. Subject has been diagnosed with osteoporosis as defined as a DXA t-score >-2.5.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
to measure the subject's pain, disability and activity level restrictions within the last week. | to measure change from pre-op (baseline) at specified intervals up to 24 months post-op
  The FFI, Foot Function Index is a validated self-administered scoring system designed to measure the subject's pain, disability and activity levels within the past week. Possible scores range from 0-100 with a lower score representing less pain, greater function and less restricted ambulation.

SECONDARY OUTCOMES:
Radiographic Evaluation | to measure change from pre-op to post-op at intervals up to 24 months postoperatively.
  Standard AP and lateral and oblique x-rays will be obtained at pre-operatively, and at 6 weeks, 3, 6, 12 and 24 months postoperatively. Any standard of care image can be performed 30 days prior to consenting.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lee, M.D., Principal Investigator — Orthopedic Foot and Ankle Center
Locations (1):
- Orthopaedic Foot and Ankle Center, Columbus, Ohio, United States